CLINICAL TRIAL: NCT07334639
Title: Metabolic Changes Associated With Weight Gain After Treatment of Achalasia
Status: Not yet recruiting | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Daniel Cohen, Gastroenterologist, Assaf-Harofeh Medical Center
Other Study IDs: 0290-25-ASF
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Achalasia, Esophageal
Keywords: achalasia; weight gain; obesity; metabolic syndrome; hepatic steatosis
MeSH Terms: conditions — Esophageal Achalasia; Weight Gain; Obesity; Metabolic Syndrome; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Achalasia patients: Patients with achalasia who undergoing treatment with either per oral endoscopic myotomy (POEM) or laparoscopic Heller myotomy (LHM). Each participant's metabolic status will be evaluated at the time of treatment and one year later.

SUMMARY:
This goal of the study is to assess the effect of weight gain in patients with achalasia after they are treated. The main question to be answered is if weight gain after achalasia treatment is associated with worsening metabolic status. Patients will be compared between their baseline status at the time of treatment and 1 year after treatment. Participants will have metabolic tests performed at these 2 times including blood tests.

DETAILED DESCRIPTION:
Background Achalasia is a disease characterized by the loss of the myenteric neurons that coordinate esophageal peristalsis and lower esophageal sphincter (LES) relaxation.1 As a result, there is aperistalsis of the esophagus and impaired LES relaxation after deglutition. The primary symptoms are dysphagia, regurgitation, and chest pain.

Weight loss is also common.2 Studies have shown weight loss occurring in between 35-69% of achalasia patients.3,4 One study reported that patients with Type II Achalasia were more likely to have weight loss than the other subtypes.5 Studies have also shown that patients with achalasia, even when not underweight, are at risk of malnutrition.6 Recently, studies have begun assessing the weight gain that occurs after successful treatment of achalasia.7-10 These studies have evaluated achalasia patients after laparoscopic Heller myotomy (LHM),7 peroral endoscopic myotomy (POEM),8,9 or a combination of treatment modalities.10 They have consistently shown significant weight gain after treatment, with many patients becoming overweight or obese.

However, the impact of this weight gain has not been objectively evaluated. Thus, to our knowledge, no studies have evaluated the cardiovascular or metabolic effects of this post-treatment weight gain.

Goals Therefore, we aim to evaluate the metabolic effects of post-treatment weight gain in in a cohort of achalasia patients undergoing treatment by assessing the relationship between weight gain and glycemic control, cholesterol levels, blood pressure, and hepatic steatosis.

Methods A prospective pilot study will be performed at both Shamir Medical Center and Hadassah Medical Center. All adult patients diagnosed with achalasia and undergoing either POEM or LHM for treatment of achalasia will be included.

The cases of achalasia will be reviewed thoroughly for demographic, clinical, laboratory, and manometric information.

Additionally, prior to POEM, the patient will be evaluated for:

* height, weight, and BMI;
* resting blood pressure;
* laboratory data including fasting glucose, Hgb A1c level, cholesterol panel, triglycerides, and liver function tests;
* Fibroscan (to measure hepatic steatosis and fibrosis).
* Eckhardt score
* Waist circumference
* Body fat percentage POEM or LHM will then be performed as indicated for achalasia treatment. One year after treatment, the initial testing will be repeated (including weight, blood pressure, fasting laboratory data, waist circumference, body fat percentage, and Fibroscan).

Statistical analyses Each patient's follow-up results will be compared to their pre-treatment results. Outcomes will include changes in levels of hepatic steatosis, waist circumference, body fat percentage, fasting glucose, Hgb A1c, cholesterol, liver function tests, and triglycerides compared to baseline, and the relationship in these changes to any weight gained. The primary outcome will be the change in hepatic steatosis on Fibroscan testing.

Continuous variables with a normal distribution will be reported as mean with standard deviation (SD), while those with a skewed distribution will be reported as median with interquartile range (IQR). Comparisons of categorical variables will be performed using the Chi-square test and Fisher's Exact test. Comparisons involving continuous variables will be performed using the Mann-Whitney U test. For all statistical calculations, a p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Proven achalasia
* Undergoing LHM or POEM for treatment

Exclusion Criteria:

* Under age 18
* Does no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with achalasia and undergoing therapy with either POEM or LHM
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Increase in Hepatic steatosis | 1 year
  The degree of hepatic steatosis assessed on FibroScan at baseline compared to 1 year later

SECONDARY OUTCOMES:
fasting glucose | 1 year
  Change in fasting glucose between baseline and 1 year later
Hgb A1c | 1 year
  Change in Hgb A1c level between baseline and 1 year later
Cholesterol | 1 year
  Change in cholesterol between baseline and 1 year later
Triglycerides | 1 year
  Change in triglycerides between baseline and 1 year later
Weight | 1 year
  Change in weight between baseline and 1 year later
waist circumference | 1 year
  Change in waist circumference between baseline and 1 year later
Body fat | 1 year
  Change in body fat percentage between baseline and 1 year later
LFTs | 1 year
  Change in liver function tests between baseline and 1 year later
Blood pressure | 1 year
  Change in resting blood pressure between baseline and 1 year later. Both the systolic and diastolic values will be assessed.
Eckhardt score | 1 year
  Change in Eckhardt score between baseline and 1 year later. The Eckhardt score goes from 0 to 12 with higher numbers meaning more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Shamir Medical Center, Ẕerifin

IPD SHARING:
Plan to Share IPD: No
The confidential information will only be used for this study.

REFERENCES:
- [Background] Patel DA, Vaezi MF. Achalasia and Nutrition: Is it Simple Physics or Biology. Pract Gastro. 2016 Nov;40(11):42-48.
- [Background] Pandolfino JE, Gawron AJ. Achalasia: a systematic review. JAMA. 2015 May 12;313(18):1841-52. doi: 10.1001/jama.2015.2996. PMID 25965233